CLINICAL TRIAL: NCT01515904
Title: Evaluation of the SickKids Team Obesity Management Program (STOMP)
Brief Title: Evaluation of the SickKids Team Obesity Management Program
Acronym: STOMP
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jill Hamilton, Staff Endocrinologist, The Hospital for Sick Children
Other Study IDs: 1000025502
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Obesity
Keywords: obesity management; adolescents; body mass index; treatment outcomes; program evaluation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Approximately 50% of attendees choose not to book into the STOMP program, for reasons including difficulty attending the frequent appointments due to distance or inability to leave work early. This population will serve as the control group for the evaluation. Control participants will be recruited from the community through posters in the hospital
- STOMP: 12-17 yrs. Patients in the program have severe complex obesity defined as children and youth who have a BMI >95th %ile for their age and gender in addition to one of the following: at least one significant obesity-related co-morbidity requiring specialty care (e.g. type 2 diabetes), other co-existing chronic illness impacted by obesity (e.g. CNS tumor, post-organ transplant), or a BMI ≥99th percentile for their age and gender
  Interventions: Behavioral: STOMP Clinic

INTERVENTIONS:
Behavioral: STOMP Clinic — A new interdisciplinary clinic (STOMP) was created to provide care for children and adolescents with severe 'complex' obesity. As part of the program, a subset of adolescents undergo bariatric surgery. The core elements include an interdisciplinary team, frequent visits, individualized care plans for medically-complex adolescents) and building on other aspects, such as increased psychosocial intervention; involvement of a "key worker" (nurse practitioner) to support families; provision of continuity of care with other health providers in all settings, community services and schools; a more diverse patient population; and group support sessions.
  Groups: STOMP

SUMMARY:
In January 2010 a new interdisciplinary clinic (STOMP) was created to provide care for children and adolescents with severe 'complex' obesity. As part of the program, a subset of adolescents undergo bariatric surgery. There is a paucity of literature evaluating outcomes of children and adolescents participating in a 'clinical' setting and even fewer reports of outcomes of severely obese pediatric patients. Previously, the investigators evaluated clinical outcomes of children with craniopharyngioma and hypothalamic obesity attending an outpatient interdisciplinary program at SickKids (The Comprehensive Care Clinic for Children with Central Tumours) and found significant benefit to those attending, including reduction of weight gain (or weight loss), improved psychosocial functioning, and increased care satisfaction. STOMP is a natural extension of this program, incorporating some core elements (e.g., interdisciplinary team, frequent visits, individualized care plans for medically-complex adolescents) and building on other aspects, such as increased psychosocial intervention; involvement of a "key worker" (nurse practitioner) to support families; provision of continuity of care with other health providers in all settings, community services and schools; a more diverse patient population; and group support sessions. Evaluation of the outcomes of this clinic is needed to inform best practice for children and adolescents with severe complex obesity

DETAILED DESCRIPTION:
The primary objective is to conduct an evaluation of the STOMP clinic as a model of care with a specific focus on: (i) patient outcomes (anthropometric, metabolic, and psychosocial); and (ii) care coordination and care satisfaction.

Patient outcomes will be compared against baseline evaluation data over time, and to a control group of patients not enrolled in the program, but who expressed interest in the program and were unable to attend.

ELIGIBILITY:
Inclusion Criteria:

* All patients enrolled in the STOMP program are eligible to participate in the study.
* Control participants must be between 12-18 years of age with a BMI >95th percentile for age.

Exclusion Criteria:

- Control participants cannot be enrolled in the STOMP program.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: STOMP Group:12-17 yrs. Patients in the program have severe complex obesity defined as children and youth who have a BMI >95th %ile for their age and gender in addition to one of the following: at least one significant obesity-related co-morbidity requiring specialty care (e.g. type 2 diabetes), other co-existing chronic illness impacted by obesity (e.g. CNS tumor, post-organ transplant), or a BMI ≥99th percentile for their age and gender Control: Approximately 50% of attendees choose not to book into the program, for reasons including difficulty attending the frequent appointments due to distance or inability to leave work early. This population will serve as the control group for the evaluation. Control participants will be recruited from the community through posters in the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-04 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index | Baseline
  BMI will be measured at Baseline and 12 months after treatment to evaluate change
Body Mass Index | 12 months
  BMI will be measured at Baseline and 12 months after treatment to evaluate change

SECONDARY OUTCOMES:
Systolic and Diastolic Blood Pressure | Baseline, 12 months
  Systolic and Diastolic Blood Pressure will be measured at Baseline and 12 months after treatment to evaluate change
Lipid profile | Baseline and 12 months
  The lipid profile (including total cholesterol, LDL cholesterol, HDL cholesterol, non-HDL cholesterol and triglycerides) will be measured at Baseline and 12 months after treatment to evaluate change
Glycemic control and Insulin resistance | Baseline and 12 months
  Glycemic control will be measured by HbA1c values and insulin resitance will be assed by HOMA-IR
Health and weight-related quality of life | Baseline and 12 months
  This outcome measure will be assessed by the Pediatric Quality of Life Inventory (PedsQL)) and the impact of Weight on Quality of Life (IWQOL)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Hamilton, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada